CLINICAL TRIAL: NCT07028502
Title: A Comparison of Two Different Transseptal Puncture Strategies Without Fluoroscopy Guidance
Acronym: TSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202209049RIPA
Record Dates: First submitted 2025-04-27; First posted 2025-06-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Ablation; Trans-septal puncture (TSP); Zero-fluoroscopy; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echocardiography (Active Comparator): The movement of the puncture needle was monitored using intracardiac echocardiography rather than fluoroscopy. All other steps followed the conventional approach.
  Interventions: Procedure: J Wire
- 3D mapping system (Experimental): Guided by the ablation catheter image on the 3D mapping system, the long sheath was advanced to the puncture site and then exchanged for a puncture needle. The entire procedure was monitored with intracardiac echocardiography.
  Interventions: Procedure: 3D mapping system

INTERVENTIONS:
Procedure: J Wire — The movement of the puncture needle was monitored using intracardiac echocardiography rather than fluoroscopy. All other steps followed the conventional approach.
  Arms: Echocardiography
Procedure: 3D mapping system — Guided by the ablation catheter image on the 3D mapping system, the long sheath was advanced to the puncture site and then exchanged for a puncture needle. The entire procedure was monitored with intracardiac echocardiography.
  Other Names: Vizigo set
  Arms: 3D mapping system

SUMMARY:
Zero-fluoroscopy is the dream of all interventionists, and as low as reasonably achievable (ALARA) is the goal the investigators can manage at this moment. Trans-septal puncture (TSP) is the most pivotal step in the ablation procedure for left heart procedure, including atrial fibrillation ablation, and it is the only step that still needs fluoroscopy in the era of 3D electroanatomical map. With the incorporation of intracardiac echocardiography (ICE), the dream of zerofluoroscopy can be achieved.

Because the imaging offered by fluoroscopy or ICE is so different in terms of the advantages and shortages, the best TSP protocols might be different. Currently, in the literature, two techniques are commonly referred. However, no comparison has been made between these two techniques. Therefore, this study is to compare the safety and efficiency of these two techniques, also to observe the transition of a senior EP doctor who has been experienced in fluoroscopy-guided TSP, hoping to establish the learning curve for future reference of zerofluoroscopy promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with paroxysmal or persistent AF and are scheduled to undergo at least but not limited to pulmonary vein (PV) isolation.
2. Patients who are willing to sign the informed consent.

Exclusion Criteria:

1. The patients need right atrial mapping and/or ablation before TSP.
2. The women who is pregnant.
3. Informed consent could not be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Total TSP time | Perioperative
  Time duration from femoral venous access to the completion of both the first and second transseptal puncture (TSP).
  Unit of Measure: Minutes
Fluoroscopy usage and radiation dose | during the procedure
  Whether fluoroscopy was used during the procedure and the corresponding radiation dose recorded if applicable.
Incidence of procedural complications | up to 12 weeks
  Occurrence of major complications during the procedure, including pericardial effusion, cardiac tamponade, stroke, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospita, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No